CLINICAL TRIAL: NCT03890146
Title: Concordance of Capillary Blood Biological Samples Analyzed in Delocalized Biology With Conventional Venous Biological Blood Samples Analyzed at the Biology Laboratory
Brief Title: Concordance of Capillary Blood Biological Samples With Conventional Venousbiological Blood Samples.
Acronym: CAPIVEIN
Status: Terminated | Type: Observational
Why Stopped: we submitted an amendment. The study was stopped because this amendment raised the complexity of the study.
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 2018-A01880-55
Record Dates: First submitted 2019-02-18; First posted 2019-03-26 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Biochemical Dysfunction
Keywords: intensive care; capillary sampling; veinous sampling; natremia; kalaemia; Chloremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intensive care patients: patient hospitalised in intensive care unit veinous and capillary ponction

SUMMARY:
The main objectives are to evaluate the concordance between the results of natremia, kalaemia and blood sugar levels obtained 1) by capillary puncture, analysed on a delocalized resuscitation machine GEM 4000 (Werfen) and 2) by venous sampling, analysed on the machine of the standard biology laboratory Gen. 2 COBAS (Roche).

DETAILED DESCRIPTION:
The completion of a biological test suits a succession of codified steps:

* Medical prescription
* The pre-analytic phase (preparation of the material, completion of the sample, transport of the sample and preparation of it)
* The analytical phase
* The post-analytic phase (validation of the result obtained and the dissemination of it to the prescriber, usually the clinician, who is then able to make a medical decision) This succession of steps involves, as part of a classical journey, many stakeholders (doctors, nurses, couriers, laboratory technicians, medical biologists) in different places.

Outsourced biology (care test point, POCT) refers to the analysis of biological samples outside the central laboratory. The sample is most often carried out, transported and analyzed by the same person on a machine near the patient or in the service and therefore in the absence of direct control of a specialized laboratory technician or a medical biologist, who remains however responsible for good practice, maintenance of the device and validity of the results.

The completion of biological examinations is regulated by differents Articles. The outsourced biology (ADBD) sampling analysis can be carried out in the hospital, in most departments, and also outside the hospital (pharmacies, city offices or even in the patient's own home). On portable devices, usually highly specialized, and these fixed allowing a greater diversity of tests.

Its development is booming with annual growth estimated in 2006 at 15.5% in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18
* Affiliate or beneficiary of a social security scheme
* Express consent to participate in the study

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Patient not communicating
* Pregnant or breastfeeding woman
* Peripheral edema (taking more than 5 Kg since entering the service)
* Patient in shock (mean arterial pressure < 65 mmHg or continuous catecholamine administration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized in the intensive care unit for any reason
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
concordance between capillary and veinous sampling for natremia result | 1 hour
  The concordance between the biological results obtained by capillary puncture analysed on the GEM 4000 resuscitation machine (Werfen), and the biological results by venous sampling analysed in the standard biology laboratory on the Gen. 2 COBAS machine (Roche) for natremia
concordance between capillary and veinous sampling for kalemia result | 1 hour
  The concordance between the biological results obtained by capillary puncture analysed on the GEM 4000 resuscitation machine (Werfen), and the biological results by venous sampling analysed in the standard biology laboratory on the Gen. 2 COBAS machine (Roche) for kalemia
concordance between capillary and veinous sampling for chloremiaresult | 1 hour
  The concordance between the biological results obtained by capillary puncture analysed on the GEM 4000 resuscitation machine (Werfen), and the biological results by venous sampling analysed in the standard biology laboratory on the Gen. 2 COBAS machine (Roche) for chloremia

CONTACTS AND LOCATIONS:
Overall Officials: Nefeli Nasika, Principal Investigator — Fonadtion Afolphe Rothschild
Locations (1):
- France, Paris, France